CLINICAL TRIAL: NCT04611516
Title: The Ear-Nose-Throat (ENT) Prospective International Cohort of PCD Patients (EPIC-PCD)
Acronym: EPIC-PCD
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Bicetre Hospital (Other); Centre Hospitalier Intercommunal Creteil (Other); University Hospital Southampton NHS Foundation Trust (Other); Universitaire Ziekenhuizen KU Leuven (Other); Amsterdam UMC, location VUmc (Other); University of Cyprus (Other); Hacettepe University (Other); Marmara University (Other); Hospital Universitario La Fe (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC-PCD
Record Dates: First submitted 2020-10-08; First posted 2020-11-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Ear-Nose-Throat (ENT) Prospective International Cohort of patients with Primary Ciliary Dyskinesia (EPIC-PCD) is a prospective observational clinical cohort study, set up as a multinational multi-centre study. It is embedded into routine patient care of participating reference centres for PCD and patients keep being managed according to local procedures and guidelines.

DETAILED DESCRIPTION:
The EPICD-PCD is hosted at the Institute of Social and Preventive Medicine (ISPM) at the University of Bern, Switzerland. Research is performed in close collaboration with all data contributors. This study aims to characterise ENT disease in PCD patients and its association with lower respiratory disease, and to identify determinants of its prognosis.

The investigators aim to:

1. Assess the prevalence and severity of sinonasal and otologic symptoms and the frequency and range of signs and physiological findings assessed during standardised ENT physical examination, and describe differences by age;
2. Study the association of sinonasal and otologic disease with lower respiratory disease in PCD patients;
3. Identify determinants of disease course and prognosis of sinonasal and otologic disease in PCD patients
4. Study management practices and identify determinants that inform them.

Study design:

The EPIC-PCD is a prospective observational clinical cohort study, set up as a multinational multi-centre study. It is embedded into routine patient care of participating reference centres for PCD and patients will keep being managed according to local procedures and guidelines.

Patients with PCD are followed regularly at each centre, at 3-month to 6-month intervals. Each patient undergoes a detailed ENT sinonasal and otologic examination by ENT specialists, at minimum once a year, during a programmed follow-up visit. Additional ENT examinations are performed if indicated during in-between follow-up visits. Patients will not be subjected to additional invasive measurements solely for the purposes of the study.

What information is collected:

The study collect clinical data from patients assessment at regular consultations at the outpatient clinics.

For the collection of clinical data, participating centres will use FOLLOW-PCD, a disease-specific form for standardised prospective data collection during routine clinical follow-up of PCD patients.

Study database:

The EPIC-PCD database is web-based, using the Research Electronic Data Capture (REDCap) platform developed at Vanderbilt University. REDCap is widely used in academic research and allows data entry and extraction in various formats.

How to participate:

Centres that wish to participate to the project and contribute data can contact the EPIC-PCD managing centre to sign a data delivery agreement. They then will receive a password to access the online software REDCap and they will be able to enter their data directly. They can also upload follow-up data or add additional patients at a later time point.

Funding:

The setting up of the EPIC-PCD (salaries, consumables and equipment) was funded by the Swiss National Science Foundation. Data collection and management at each site was funded according to local arrangements. Most participating researchers and data contributors participate in the European Respiratory Society Clinical Research collaboration "Better Evidence to Advance Therapeutic options for PCD" (BEAT-PCD) (https://beat-pcd.squarespace.com/). Infrastructure is provided for free by the University of Bern, where the data are pooled and stored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCD (clinical and test certified)
* Patient must undergo an ENT examination minimum once a year as part of their clinical follow-up

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages diagnosed with PCD, followed in a collaborating PCD centre
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Sinonasal symptoms and signs | at baseline
  Prevalence of reported clinical symptoms at different age groups, including rhinitis, sinusitis, snoring
Course of sinonasal symptoms and signs (year 1) | at 12 months from recruitment
  Change from baseline prevalence of reported clinical symptoms at different age groups, including rhinitis, sinusitis, snoring, at 12 months
Course of sinonasal symptoms and signs (year 2) | at 24 months from recruitment
  Change from baseline prevalence of reported clinical symptoms at different age groups, including rhinitis, sinusitis, snoring, at 24 months
Otological symptoms and signs | at baseline
  Prevalence of reported clinical symptoms at different age groups, including ear pain, hearing problems, ear discharge
Course of otological symptoms and signs (year 1) | at 12 months from recruitment
  Change from baseline prevalence of reported clinical symptoms at different age groups, including ear pain, hearing problems, ear discharge, at 12 months
Course of otological symptoms and signs (year 2) | at 24 months from recruitment
  Change from baseline prevalence of reported clinical symptoms at different age groups, including ear pain, hearing problems, ear discharge, at 24 months
Nasal endoscopy (description of nasal mucosa) | at baseline
  Description of nasal mucosa as seen via nasal endoscopy examination
Nasal endoscopy (changes of nasal mucosa at year 1) | at 12 months from recruitment
  Changes in nasal mucosa from baseline as seen via nasal endoscopy examination at 12 months
Nasal endoscopy (changes of nasal mucosa at year 2) | at 24 months from recruitment
  Changes in nasal mucosa from baseline as seen via nasal endoscopy examination at 24 months
Nasal endoscopy (nasal polyps) | at baseline
  Prevalence of nasal polyps at baseline
Nasal endoscopy (nasal polyps at year 1) | at 12 months from recruitment
  Changes in prevalence of nasal polyps from baseline to 12 months
Nasal endoscopy (nasal polyps at year 2) | at 24 months from recruitment
  Changes in prevalence of nasal polyps from baseline to 24 months
Sinonasal examination (Lidholdt score) | at baseline
  Lidholdt score at baseline
Sinonasal examination (Lidholdt score at year 1) | at 12 months from recruitment
  Changes in Lidholdt score from baseline to 12 months
Sinonasal examination (Lidholdt score at year 2) | at 24 months from recruitment
  Changes in Lidholdt score from baseline to 24 months
Ear examination (ear discharge) | at baseline
  Prevalence of ear discharge at baseline
Ear examination (ear discharge at year 1) | at 12 months from recruitment
  Changes in prevalence of ear discharge from baseline to 12 months
Ear examination (ear discharge at year 2) | at 24 months from recruitment
  Changes in prevalence of ear discharge from baseline to 24 months
Otoscopy (description of the tympanic membrane) | at baseline
  Description of tympanic membrane as seen via otoscopy examination
Otoscopy (description of the tympanic membrane at year 1) | at 12 months from recruitment
  Changes in the tympanic membrane from baseline to 12 months as seen via otoscopy examination
Otoscopy (description of the tympanic membrane at year 2) | at 24 months from recruitment
  Changes in the tympanic membrane from baseline to 24 months as seen via otoscopy examination
Tympanometry | at baseline
  Results of tympanometry (tympanogram type for both ears) at baseline
Tympanometry (at year 1) | at 12 months from recruitment
  Changes in tympanogram (for both ears) from baseline to 12 months
Tympanometry (at year 2) | at 24 months from recruitment
  Changes in tympanogram (for both ears) from baseline to 24 months
Audiometry | at baseline
  Results of audiometry: type of audiometry and results based on WHO hearing loss grades (for both ears)
Audiometry (at year 1) | at 12 months from recruitment
  Changes in audiometry results from baseline to 12 months
Audiometry (at year 2) | at 24 months from recruitment
  Changes in audiometry results from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Myrofora Goutaki, MD-PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Not all participating centres have ethical approval to share IPD to external researchers.
  Researchers wanting to use the dataset can propose a research topic and draft a concept sheet describing the planned analyses and publication. All concept sheets have to be approved by all participating centres contributing data to the proposed analysis under question. After the participating centres agree to contribute their data and sign a publication agreement, the EPIC-PCD managing centre (University of Bern) will prepare a partial dataset for the proposed analysis and will work closely with the lead researchers offering methodological input and support. In case additional data is collected to complete the partial dataset for a specific project, this will be added to the EPIC-PCD dataset to enrich it after each project.

REFERENCES:
- [Derived] Goutaki M, Lam YT, Alexandru M, Anagiotos A, Armengot M, Bequignon E, Boon M, Burgess A, Coste A, Emiralioglu N, Erdem E, Haarman EG, Harris A, Hool SL, Karadag B, Kim S, Latzin P, Lorent N, Ozcelik U, Reula A, Roehmel J, van Gogh C, Yiallouros P, Zappe SM; EPIC-PCD team; Papon JF. Study protocol: the ear-nose-throat (ENT) prospective international cohort of patients with primary ciliary dyskinesia (EPIC-PCD). BMJ Open. 2021 Oct 11;11(10):e051433. doi: 10.1136/bmjopen-2021-051433. PMID 34635525